CLINICAL TRIAL: NCT07144085
Title: Application of ⁶⁸Ga-FXX489 (NNS309) PET/CT Imaging in Diagnosis of Tumor Diseases.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yi Tian (Other)
Responsible Party: Sponsor-Investigator, Yi Tian, The Master's Degree Candidate of the Department of Nuclear Medicine, The First Affiliated Hospital of China Medical University, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: [2025]670
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Tumor; Metastatic Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor population (Experimental): PET imaging will begin 30 +/-10 minutes, 60 +/-15 minutes and 120 +/-20 minutes after injection of 68Ga-FXX489 or 68Ga-FAP-2286 or 18F-FDG.
  Interventions: Drug: 68Ga-FXX489; Procedure: Positron Emission Tomography (PET) imaging; Drug: Gallium-68 labelled (68Ga-) FAP-2286

INTERVENTIONS:
Drug: 68Ga-FXX489 — The dose will be 3 to 8 millicurie (mCi) +/- 10% given intravenously at a single time prior to imaging.
Procedure: Positron Emission Tomography (PET) imaging — Participants will be scanned for approximately 30 to 45 minutes.
Drug: Gallium-68 labelled (68Ga-) FAP-2286 — The dose will be 3 to 8 millicurie (mCi) +/- 10% given intravenously at a single time prior to imaging.

SUMMARY:
A new radiotracer, 68Ga-FXX489 (NNS309), has been developed for tracking fibroblast activation protein (FAP) and visualizing the tumor stroma. The purpose of the study is to explore the diagnostic value of 68Ga-FXX489 (NNS309) PET/CT imaging in oncological diseases, to assess its safety, imaging characteristics, and biodistribution after administration.

DETAILED DESCRIPTION:
Initially the investigator(s) will focus on imaging pancreatic cancer, lung cancer, breast cancer, gastric cancer, colorectal cancer.

STUDY AIMS

1. Determine the dosimetry for gallium-68 labelled 68Ga- FXX489(NNS309).
2. Evaluate the uptake and retention of radiotracer in a variety of solid tumors with 68Ga- FXX489(NNS309).
3. Evaluate the ability of FAP-2286 to detect metastatic disease. PRIMARY OBJECTIVES

1.Safety of 68Ga- FXX489(NNS309). 2.determine the organ dosimetry of 68Ga- FXX489(NNS309). 3.To assess the feasibility of detecting tumor uptake using FXX489(NNS309). 4.To determine the feasibility of detecting metastatic disease using FXX489(NNS309).

EXPLORATORY OBJECTIVES

1. Determine impact of administered dose of FXX489(NNS309) on image quality.
2. Compare the feasibility of detecting tumor uptake using FXX489(NNS309) and FAP-2286 .

A repeat radiolabeled FXX489(NNS309) PET may be obtained after initiation of subsequent treatment in order to evaluate changes in PET uptake due to treatment effect. Patients will be followed for up to 3 days after the injection of radiolabeled ligand for evaluation of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a high suspicion of oncological diseases.
2. Age: 18-80 years, no gender restriction, able to express themselves independently, and willing to participate in this study with a signed informed consent form.

Exclusion Criteria:

1. Failure to sign the informed consent form.
2. Severe visual or auditory impairment, cognitive disorders, or patients with claustrophobia who cannot communicate effectively.
3. Severe cardiac dysfunction, cardiac function class III-IV.
4. Renal failure (serum creatinine level > 1.2 mg/dl).
5. Allergy to alcohol.
6. Use of drugs within 1 week prior to the examination that can cause a disulfiram-like reaction with alcohol, such as penicillins, cephalosporins, or cefotetan.
7. Known pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Count of participants with treatment-emergent adverse events | Up to 3 days
  The frequency and severity of treatment emergent adverse events following FXX489(NNS306) injection will be descriptively reported as classified and graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Proportion of radiation-absorbed doses of radiolabeled FAP-2286. | Up to 3 days
  Volumes of interest of 68Ga- will be drawn around regions identified on the scans, including the liver, spleen, kidneys, urinary bladder, the central sacrum (for hematopoietic marrow) and whole body. Data will be fitted using the Simulation, Analysis, and Modeling Software II (SAAM II) software. Time integrals of activity will be entered into the Organ Level INternal Dose Assessment/EXponential Modeling (OLINDA/EXM) software, using the reference adult model. The results from all patients enrolled will be combined to allow the calculation of mean, standard deviation (SD), and range of radiation-absorbed doses to individual organs
Standardized Uptake Values (SUVs) | Up to 3 days
  The maximum Standardized Uptake Value (SUVmax) will be calculated for up to five lesions in each patient, with mediastinal blood pool being used as background activity.
Tumor-to-background (TBR) Ratio | Up to 3 days
  TBR ratios will be calculated for up to five lesions in each patient, with mediastinal blood pool being used as background activity. The median and range of the measured TBRs will be reported across all RECIST measurable lesions as a table broken down by location (organ metastases, nodal metastases and bone metastases).
Proportion of positive lesions on FXX489(NNS306) PET | Up to 3 days
  Conventional imaging will be reviewed in conjunction with the FXX489(NNS306) PET images. Lesions will be characterized as positive on FXX489(NNS306) PET if uptake is greater than 1.5 times higher than mediastinal blood pool and uptake cannot be attributed to physiologic or inflammatory reasons. Conventional imaging will be interpreted as positive by each lesion if the short axis dimension of lymph nodes is greater than 1 centimeter (cm), and organ metastases measure greater than 1 cm in long axis. The gold standard will be the combination of conventional imaging and FXX489(NNS306) PET in combination with clinical follow-up and histopathology (if available). The number of lesions detected by each modality will be compared and sensitivity will be computed. Since this is a proof-of-concept study, it is not powered for the test of agreement. Nevertheless, the agreement will be tested using McNemar's test.

CONTACTS AND LOCATIONS:
Overall Officials: Xuena Li, Study Director — Department of Nuclear Medicine, The First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No